CLINICAL TRIAL: NCT03917901
Title: Computer-Delivered Intervention for Individuals With Obesity and Elevated Anxiety Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Brooke Kauffman, Principal Investigator, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001405
Record Dates: First submitted 2019-04-13; First posted 2019-04-17 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Anxiety Sensitivity; Eating; Physical Activity
Keywords: Anxiety Disorders; Depression; Anxiety Sensitivity; Obesity; Eating; Physical Activity; Exercise
MeSH Terms: conditions — Obesity; Motor Activity; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: If participant meets eligibility criteria, the participant will be randomly assigned to complete a one-session computer-delivered intervention: either (1) anxiety sensitivity reduction treatment or (2) health information control.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anxiety Sensitivity Training (Experimental): The Anxiety Sensitivity training (AST) will provide: (1) psychoeducation on anxiety sensitivity and its consequences, (2) psychoeducation on the relationship between anxiety sensitivity and obesity-related health behavior correlates, and (3) concrete, evidenced-based strategies to reduce anxiety sensitivity.
  Interventions: Other: Anxiety Sensitivity Training
- Health Control (Placebo Comparator): The Health Control (HC) will cover general health care, such as information on wearing sunscreen and regular attendance to doctor appointments. The HC will not provide any recommendations or education on mood, dietary, or physical habits.
  Interventions: Other: Health Control

INTERVENTIONS:
Other: Anxiety Sensitivity Training — Computerized Single-Session Anxiety Sensitivity Reduction Program
  Arms: Anxiety Sensitivity Training
Other: Health Control — Computerized Single-Session Health Information Control
  Arms: Health Control

SUMMARY:
The proposed study will design and evaluate a computerized-delivered single-session anxiety sensitivity reduction program (i.e., Anxiety Sensitivity Training; AST). The AST will be designed to achieve three primary aims: (1) provide psycho-educational information on AS and its consequences, (2) present psycho-educational information on the relationship between AS and obesity-related health behavior correlates, and (3) offer concrete, evidence-based strategies to facilitate motivation to change their obesity-related lifestyle behaviors.

DETAILED DESCRIPTION:
The primary goal of the research study is to investigate the efficacy of a brief, computer-delivered transdiagnostic intervention that addresses anxiety sensitivity to reduce emotional eating, eating expectancies, food cravings, binge eating, perceived barriers to engage in physical activity, anxiety/depressive symptoms, severity of daily fatigue and increase perceived benefits to engage in physical activity, exercise self-efficacy, willingness to use adaptive coping strategies, and perceived physical health functioning. To address this aim, the investigator's will implement a randomized controlled trial that will employ a longitudinal experimental design and involve five stages: (a) online pre-screener; (b) baseline survey consisting of a pre-intervention assessment (eligibility) and random assignment to a one-session computer-delivered intervention (Active versus Control); (c) 1-week follow-up survey; (d) 2-week follow-up survey; (e) 1-month follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index of at least 30
* Endorse elevated anxiety sensitivity defined as an ASI-3 score of 17 or greater

Exclusion Criteria:

* Any anticipated matters that would interfere with participating in the study
* Not being fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Kauffman, MA, Principal Investigator — University of Houston; Michael J Zvolensky, Ph.D., Principal Investigator — University of Houston
Locations (1):
- Anxiety and Health Research Lab, Substance Use Treatment Clinic, University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project Website — https://www.uh.edu/class/psychology/clinical-psych/research/restore/index

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anxiety Sensitivity Training | Health Control
Started | 65 | 66
1-Week Follow-up | 59 | 60
2-Week Follow-up | 62 | 57
1-Month Follow-up | 61 | 63
Completed | 65 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anxiety Sensitivity Training | Health Control | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.06 (8.90) | 31.83 (11.45) | 30.95 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 43 | 80
  Male | 28 | 23 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 42 | 38 | 80
  Race: Black or African American | 10 | 16 | 26
  Race: Asian | 5 | 4 | 9
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Other | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 65 | 66 | 131
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 38.11 (5.98) | 38.20 (5.80) | 38.15 (5.87)

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Sensitivity Index-3
Description: The Anxiety Sensitivity Index-3 is an 18-item measured that will be used to assess sensitivity to, and fear of, the potential negative consequences of anxiety-related symptoms and sensations. Items are rated on a 5-point Likert scale, ranging from 0 (Very Little) to 4 (Very Much). Scores will be calculated by summing all items (possible range = 0 -72), with lower scores indicating a better outcome.
Time Frame: Baseline,1-week, 2-week and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Sensitivity Training | Health Control
Number analyzed (Participants) | 65 | 66
score on a scale
  Baseline | 43.44 (12.27) | 43.00 (12.43)
  1-Week Follow-up: number analyzed (Participants) | 59 | 60
  1-Week Follow-up | 40.17 (14.03) | 40.69 (13.15)
  2-Week Follow-up: number analyzed (Participants) | 62 | 57
  2-Week Follow-up | 38.00 (15.13) | 37.24 (14.10)
  1-Month Follow-up: number analyzed (Participants) | 61 | 63
  1-Month Follow-up | 37.74 (16.29) | 34.25 (13.93)

2. Primary Outcome: Dutch Eating Behavior Questionnaire
Description: The Dutch Eating Behavior Questionnaire will be used to assess emotional eating. Items are rated on a 5-point Likert scale ranging from 1 (never) to 5 (very often). For the current study, the emotional eating subscale (13 items) will be used as a measure of emotional eating. The 13 items of the subscale are summed and divided by 13 to create a mean score with a range from 1-5. Lower scores on this measure indicate better outcomes.
Time Frame: Baseline,1-week, 2-week and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Sensitivity Training | Health Control
Number analyzed (Participants) | 65 | 66
score on a scale
  Baseline | 3.58 (0.91) | 3.68 (0.87)
  1-Week Follow-up: number analyzed (Participants) | 59 | 60
  1-Week Follow-up | 3.54 (1.03) | 3.59 (0.92)
  2-Week Follow-up: number analyzed (Participants) | 62 | 57
  2-Week Follow-up | 3.31 (1.08) | 3.52 (0.94)
  1-Month Follow-up: number analyzed (Participants) | 61 | 63
  1-Month Follow-up | 3.21 (1.15) | 3.35 (0.98)

3. Primary Outcome: Eating Expectancy Inventory
Description: The Eating Expectancy Inventory will be used to measure cognitive expectancies of eating. The Eating Expectancy Inventory subscale facet: eating helps manage negative affect will be used in the current study. Respondents will be asked to rate on a 7-point Likert scale the degree to which they 1 (completely disagree) to 7 (completely agree) to each item. Responses are summed for each subscale. Lower scores on the 18-item eating helps manage negative affect subscale (possible range = 18 - 126) indicate better outcomes.
Time Frame: Baseline,1-week, 2-week and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Sensitivity Training | Health Control
Number analyzed (Participants) | 65 | 66
score on a scale
  Baseline | 88.17 (22.11) | 90.06 (20.69)
  1-Week Follow-up: number analyzed (Participants) | 59 | 60
  1-Week Follow-up | 85.98 (25.89) | 89.03 (23.08)
  2-Week Follow-up: number analyzed (Participants) | 62 | 57
  2-Week Follow-up | 82.19 (26.18) | 88.30 (23.15)
  1-Month Follow-up: number analyzed (Participants) | 61 | 63
  1-Month Follow-up | 80.74 (28.71) | 87.51 (22.59)

4. Primary Outcome: Exercise Self-Efficacy
Description: Exercise self-efficacy will be assessed with a 5-item self-report assessment of one's confidence about their ability to engage in physical activity. Items are rated on a 9-point Likert-type scale that ranges from 0 (not at all confident) to 8 (extremely confident). A total score will be created by summing the 5-items with higher scores indicating a better outcome (possible range 0 - 40).
Time Frame: Baseline,1-week, 2-week and 1-month follow-up
Population: Overall number is different from analyzed number due to participants not completing select follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Sensitivity Training | Health Control
Number analyzed (Participants) | 65 | 66
score on a scale
  Baseline | 14.11 (9.31) | 16.59 (8.13)
  1-Week Follow-up: number analyzed (Participants) | 59 | 60
  1-Week Follow-up | 16.37 (9.77) | 18.06 (8.11)
  2-Week Follow-up: number analyzed (Participants) | 62 | 57
  2-Week Follow-up | 15.52 (9.14) | 17.54 (8.48)
  1-Month Follow-up: number analyzed (Participants) | 61 | 63
  1-Month Follow-up | 16.32 (9.51) | 17.20 (8.20)

ADVERSE EVENTS:
Time Frame: 1-month
Arm/Group | Anxiety Sensitivity Training | Health Control
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66
Other Adverse Events (participants affected / at risk) | 0/65 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03917901/Prot_SAP_000.pdf